CLINICAL TRIAL: NCT00392548
Title: Urinary VEGF and MMP Levels in Patients Receiving Radiation Therapy for Glioblastoma Multiforme: Prospective Determination of a Predictive Value for Recurrence
Brief Title: URINARY VEGF Levels in GBM Patients on Radiation Treatment Protocol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Radiation Therapy Oncology Group (Network)
Other Study IDs: RTOG0611
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-09

CONDITIONS: Glioblastoma
Keywords: GBM; glioblastoma; urine; VEGF; radiation; Patients must be enrolled to an RTOG GBM study that prescribes 6000 cGy of radiation therapy.
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Study of the urinary vascular endothelial growth factor (VEGF) levels in patients with glioblastoma, receiving standard therapy.

Hypothesis: that urinary VEGF levels can serve as a predictor of treatment response and survival.

DETAILED DESCRIPTION:
Measurement of urinary VEGF levels pre treatment,immediately after treatment, and 1 month after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient must be enrolled on an RTOG GBM study that prescribes 6000 cGy of radiation therapy.
* Patient must meet the eligibility requirements for the RTOG treatment study. (If the patient is deemed retrospectively ineligible for the RTOG treatment study, the patient will likewise be ineligible for this study.)
* Patient must sign a study-specific informed consent for RTOG 0611 prior to study entry.

Exclusion Criteria:

* Patient not able to receive 6000 cGy of radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2006-10; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Deborah T Blumenthal, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- tel Aviv Sourasky Medical Center, Tel Aviv, Israel